CLINICAL TRIAL: NCT00249587
Title: Medication Adherence Therapy for Opioid Abusing Pain Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Deborah Haller, Ph.D., St. Luke's-Roosevelt Hospital Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-13169-1; R01-13169-1
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2008-09

CONDITIONS: Pain; Chronic Disease; Prescription Opioid Abuse
MeSH Terms: conditions — Pain; Chronic Disease; Opioid-Related Disorders | interventions — Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Methadone plus behavioral counseling consisting of adherence, self-monitoring, and motivational interviewing
  Interventions: Drug: Methadone
- 2 (Active Comparator): Methadone plus behavioral counseling consisting of adherence
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Methadone — dosed to effect, every six hours

SUMMARY:
The purpose of this study is to develop and pilot test a combined behavioral and pharmacological intervention designed to decrease pain, functional interference, and drug abuse while increasing medication adherence.

DETAILED DESCRIPTION:
Project Pain is a Stage I behavioral therapies development project aimed at developing and pilot testing a novel intervention for patients with chronic non-malignant pain who have experienced difficulty managing prescribed opioids. The goals of the study are to: (1) develop the intervention and training materials; (2) develop therapist adherence and competence scales; (3) train therapists to deliver the intervention per the treatment protocol; and (4) pilot the intervention to assess its feasibility, acceptability and promise. The goals of the intervention are to: (1) improve adherence to prescribed opioids; (2) decrease the severity of patients' pain; and (3) improve patients' functioning and quality of life .

ELIGIBILITY:
Inclusion Criteria:

* Uninterrupted pain of at least 6 months duration
* Pain is continuous, rather than intermittent
* Pain in the severe range (VAS = 7-10) while medicated
* Poor response to non-pharmacological interventions for pain (if appropriate)
* One or more of the following pain diagnoses: (a) back/neck pain; (b) myofacial pain; (c) neuropathic pain (e.g., diabetic or AIDS neuropathy, Complex regional pain syndrome); (d) arthritic pain; (e) MS; or (f) sickle cell (must meet chronicity criteria)
* Evidence of tolerance/physiological dependence on opioid analgesics
* Current opioid use disorder (DSM-IV criteria)
* Continuous use of opioid analgesics for a minimum of 6 months prior to referral. [Note: This is consistent with minimum 6-month requirement for diagnosis of chronic pain].
* Minimum of 2 signs/symptoms of medication mismanagement identified by the Referring MD (PROBLEMS WITH PAIN MEDS checklist)

Exclusion Criteria:

* Please contact site regarding exclusion criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2000-09; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Medication compliance and unauthorized drug use | 24 weeks
Changes in pain severity and functioning | 24 weeks

SECONDARY OUTCOMES:
Satisfaction with services | 12 weeks
Therapeutic alliance | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Haller, Principal Investigator — St. Luke's Roosevelt Hosp Cntr (New York)
Locations (1):
- Behavioral Science Research Unit, New York, New York, United States

REFERENCES:
- [Background] Haller, D.L., Heckman-Stone, C. Ingersoll, K.: Drug and Alcohol Dependence. 2002; 66, S73, #270
- [Background] Wunsch, M.J., Cropsey, K.L., Haller, D.L.: Drug and Alcohol Dependence. 2002; 66, S198, #747
- [Background] Fox, S.A., Haller, D.L., Weaver, M.F.: Proceedings from CPDD 2003 Annual Meeting, Bal Harbour, Florida. #197
- [Background] Paper presented at the American Academy of Addiction Psychiatry, December, 2004